CLINICAL TRIAL: NCT02837536
Title: Horizontal vs. Vertical Positioning of the iCare Rebound Tonometer and Effects on Intraocular Pressure Readings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Robert Cizik Eye Clinic (Other)
Responsible Party: Principal Investigator, Robert Feldman, M.D., The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-16-0396
Record Dates: First submitted 2016-07-08; First posted 2016-07-19 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Horizontal iCare (Active Comparator): In the horizontal iCare arm, these patients were randomized to have their IOP measured with the iCare tonometer held in the horizontal position first and then their IOP measured with the iCare tonometer held in the vertical position.
  Interventions: Other: Horizontal iCare; Other: Vertical iCare
- Vertical iCare (Active Comparator): In the vertical iCare arm, these patients were randomized to have their IOP measured with the iCare tonometer held in the vertical position first and then their IOP measured with the iCare tonometer held in the horizontal position.
  Interventions: Other: Horizontal iCare; Other: Vertical iCare

INTERVENTIONS:
Other: Horizontal iCare — IOP of the right eye will be measured using the iCare tonometer held in the horizontal position first and then in the vertical position.
Other: Vertical iCare — IOP of the right eye will be measured using the iCare tonometer held in the vertical position first and then in the horizontal position.

SUMMARY:
The goal of this study is to evaluate the agreement between intraocular pressure (IOP) measurements taken by iCare, held in both vertical and horizontal positions. In addition, iCare measurements will be compared against pneumotonometry measurements to assess for accuracy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must be able to understand and sign and informed consent form that has been approved by an Institutional Review Board/Ethics Committee

Exclusion Criteria:

* Evidence of corneal epithelial defects or pathology affecting corneal rigidity
* Use of topical ophthalmic medications (except for artificial tears)
* History or corneal surgeries
* Any condition that would prevent or inhibit intraocular pressure measurements using iCare or pneumotonometry
* Evidence of ocular infection 30 days prior to enrollment
* Allergy to proparacaine or latex

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
IOP taken by iCare - horizontal | 1 Day
IOP taken by iCare - vertical | 1 Day
IOP taken by pneumatonometer | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Feldman, M.D., Principal Investigator — Robert Cizik Eye Clinic
Locations (1):
- Robert Cizik Eye Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No